CLINICAL TRIAL: NCT05303454
Title: Cartoons and Musical-moving Toys in Invasive Procedure Applications Reduce Pain and Fear Levels of Children: A Randomized Controlled Study
Brief Title: Cartoons and Musical-moving Toys in Invasive Procedure Applications Reduce Pain and Fear Levels of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.O.oı.OO/36
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pediatric Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cartoons (Experimental): Reduce Pain and Fear Levels of Children
  Interventions: Behavioral: Cartoons
- Musical-moving Toys (Experimental): Reduce Pain and Fear Levels of Children
  Interventions: Behavioral: musical-moving toys
- CONTROL (No Intervention): NOT Reduce Pain and Fear Levels of Children

INTERVENTIONS:
Behavioral: Cartoons — cartoons were found to be effective in reducing children's pain and fear levels.
  Arms: Cartoons
Behavioral: musical-moving toys — musical-moving toys were found to be effective in reducing children's pain and fear levels.
  Arms: Musical-moving Toys

SUMMARY:
Aim: The aim of this study is to determine the effect of the cartoon and musical-moving toy watched in the invasive procedure application on the pain and fear level of children.

Material and Method: The research was carried out as a randomized controlled experiment in Atatürk University Health Research and Application Center Pediatric Emergency Service between March 2021 and February 2022. The population of the study consisted of children between the ages of 3 and 6 who came for treatment at the specified hospital. The sample of the research; 40 cartoons, 40 musical-moving toys, 40 control group, totally 120 children who applied to the pediatric emergency service between June 2021 and January 2022 and met the research criteria and volunteered to participate in the research. Data collection tools were collected through face-to-face interviews with "Survey Form", "Wong-Baker Faces Pain Rating Scale (WBS)" and "Child Fear Scale (CFS)". In the research, "cartoon" and "musical-moving toy" were used as intervention tools.

DETAILED DESCRIPTION:
Aim: The aim of this study is to determine the effect of the cartoon and musical-moving toy watched in the invasive procedure application on the pain and fear level of children.

Material and Method: The research was carried out as a randomized controlled experiment in Atatürk University Health Research and Application Center Pediatric Emergency Service between March 2021 and February 2022. There is one intervention room in the Pediatric Emergency Service. There are blood collection stretcher, vascular access-bleeding materials (intraket, cotton, 70% alcohol, tourniquet, plaster, injector, blood tubes, etc.) in this room.The population of the study consisted of children between the ages of 3 and 6 who came for treatment at the specified hospital. In order to ensure randomization, the children who met the criteria were included in the control group in the first week, the children in the second week were included in the cartoon group, and the children in the third week were included in the musical-moving toy group, and this cycle was continued until the end of the study and randomization was achieved.The sample of the research; 40 cartoons, 40 musical-moving toys, 40 control group, totally 120 children who applied to the pediatric emergency service between June 2021 and January 2022 and met the research criteria and volunteered to participate in the research. Children from 2 experimental and 2 control groups who did not want to participate in the study were excluded from the study. Prior power analysis was performed to determine the adequacy of the sample size of the study. In the power analysis, it was determined that the study was at the significance level of 0.05, at the 95% confidence interval, and the effect size was 0.551 and the power was 0.99. Data collection tools were collected through face-to-face interviews with "Survey Form", "Wong-Baker Faces Pain Rating Scale (WBS)" and "Child Fear Scale (CFS)". In the research, "cartoon" and "musical-moving toy" were used as intervention tools. Two different cartoons were used in the research, and these were the children's favorites, 'Red Fish' and 'Niloya'. Pepee is a toy suitable for the developmental characteristics of children aged three and over. The data were analyzed with the SPSS for Windows 22 package program. Ethical principles were followed in the research. The research sample is limited to pediatric patients who applied to Atatürk University Health Research and Application Center Pediatric Emergency Service between June and December 2021 and participated in the study voluntarily. Research results can be generalized to this group.

ELIGIBILITY:
Inclusion Criteria:

* between 3-6 years old,
* Does not have a chronic disease,
* Does not have a disability related to developmental areas,
* Not receiving inpatient treatment in the hospital,
* No history of sedative, analgesic or narcotic substance use within 24 hours before admission,
* Not having a febrile illness at the time of application,
* Children whose parents were with the child during the procedure were included in the study.

Exclusion Criteria:

* NOT aged between 3-6 years,
* Having a chronic illness
* Having a disability related to developmental areas,
* Receiving inpatient treatment in the hospital,
* Having a history of sedative, analgesic or narcotic substance use within 24 hours before admission,
* Having a febrile illness at the time of application,
* Children whose parents were not present during the procedure were included in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale | 8 MONTHS
  This scale is used to diagnose pain in children aged 3-18 years. In this scale, there are six facial expressions representing the increasing pain intensity from 0 to 5 from left to right. The leftmost facial expression has a smiling expression indicating a pain-free state, while the rightmost facial expression has a crying expression corresponding to the most severe pain. The child is instructed to choose the face that best expresses his or her feelings. Six facial expressions are scored between 0-5 points from left to right (0 points = very happy/no pain, 5 points = indicates the most severe pain). As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.
Child Fear Scale | 8 MONTHS
  The CLS is a scale of 0-4, showing five faces ranging from a neutral expression (0 = no concern) to the feared face (4 = severe anxiety). The child is told to choose the best facial expression that expresses his or her feelings. As the score obtained from the scale increases, the child's fear level increases.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED